CLINICAL TRIAL: NCT03225716
Title: A Phase 1/2 Study of Ulocuplumab And Ibrutinib in Symptomatic Patients With Mutated CXCR4 Waldenstrom's Macroglobulinemia
Brief Title: A Study of Ulocuplumab And Ibrutinib in Symptomatic Patients With Mutated CXCR4 Waldenstrom's Macroglobulinemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to end follow-up early
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Steven Treon, MD, PhD, MD, PhD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-235
Record Dates: First submitted 2017-06-29; First posted 2017-07-21 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2023-11

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: Waldenstrom's Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — ulocuplumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Dose level 1: Ibrutinib + Ulocuplumab 400mg Cycle 1 and 800mg Cycles 2-6 (Experimental): * Ibrutinib administered orally once daily for 48 cycles
  * Ulocuplumab administered intravenously at 400mg for Cycle 1 on Days 1, 8, 15, and 22. Ulocuplumab administered IV at 800mg for Cycles 2-6 on Days 1 and 15.
  Interventions: Drug: Ulocuplumab; Drug: Ibrutinib
- Phase 1 Dose level 2: Ibrutinib + Ulocuplumab 800mg Cycle 1 and 1200mg Cycles 2-6 (Experimental): * Ibrutinib administered orally once daily for 48 cycles
  * Ulocuplumab administered intravenously at 800mg for Cycle 1 on Days 1, 8, 15, and 22. Ulocuplumab administered IV at 1200mg for Cycles 2-6 on Days 1 and 15.
  Interventions: Drug: Ulocuplumab; Drug: Ibrutinib
- Phase 1 Dose level 3: Ibrutinib + Ulocuplumab 800mg Cycle 1 and 1600mg Cycles 2-6 (Experimental): * Ibrutinib administered orally once daily for 48 cycles
  * Ulocuplumab administered intravenously at 800mg for Cycle 1 on Days 1, 8, 15, and 22. Ulocuplumab administered IV at 1600mg for Cycles 2-6 on Days 1 and 15.
  Interventions: Drug: Ulocuplumab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Ulocuplumab — Ulocuplumab is a type of protein called an antibody that attacks CXCR4
  Other Names: BMS-936564
Drug: Ibrutinib — Ibrutinib small-molecule inhibitor of Bruton's tyrosine kinase (BTK) with potential antineoplastic activity
  Other Names: Imbruvica

SUMMARY:
This research study is studying Ulocuplumab combined with ibrutinib as a possible treatment for symptomatic Waldenstrom's Macroglobulinemia (WM).

DETAILED DESCRIPTION:
This was planned to be a Phase I/II clinical trial. A Phase I clinical trial tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied. The study was halted early and did not open the Phase II portion.

The FDA (the U.S. Food and Drug Administration) has not approved Ulocuplumab as a treatment for any disease. Ulocuplumab is a type of protein called an antibody that attacks CXCR4, a protein that is found on B-cells like WM.

The FDA (the U.S. Food and Drug Administration) has Ibrutinib as a treatment option for this disease.

Ibrutinib has been under investigation in research studies in participants with recurrent B-cell lymphoma, chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), mantle cell lymphoma (MCL), diffuse large B-cell lymphoma (DLBCL), and prolymphocytic leukemia, and WM. In a study of ibrutinib in relapsed/refractory WM patients, response rates were high and the treatment was well tolerated. In that study participants who had a CXCR4 mutation had a lower response rate to ibrutinib than those without a mutation.

In this research study, the investigators are evaluating the safety of ulocuplumab in combination with ibrutinib participants with symptomatic WM who have a CXCR4 mutation. The investigators are also evaluating how well the ulocuplumab works in combination with ibrutinib

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenstrom's Macroglobulinemia and meeting criteria for treatment using consensus panel criteria from the Second International Workshop on Waldenstrom's macroglobulinemia (Kyle et al, 2003) or have high risk disease with an serum IgM level of 6,000 mg or higher (Gustine et al, 2016).
* MYD88 and CXCR4 mutated disease (determined by Treon laboratory or molecular diagnostics laboratory).
* Measurable disease, defined as presence of serum immunoglobulin M (IgM) with a minimum IgM level of >2 times the upper limit of normal of each institution is required.
* Age ≥ 18 years
* ECOG performance status < or = 2 (see Appendix A.).
* To establish eligibility, participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,000/uL
  * Platelets ≥ 75,000/uL
  * Hemoglobin ≥ 8 g/dL
  * Total bilirubin ≤ 1.5 mg/dL or < 2 mg/dL if attributable to hepatic infiltration by neoplastic disease or Gilbert's syndrome
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional upper limit of normal
  * Creatinine ≤ 2 mg/dL
* Not on any active therapy for other malignancies with the exception of topical therapies for basal cell or squamous cell cancers of the skin.
* Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or have or will have complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) while participating in the study; and 2) for at least 28 days after discontinuation from the study. Men must agree to use a latex condom during sexual contact with a FCBP even if the participants have had a successful vasectomy. FCBP must be referred to a qualified provider of contraceptive methods if needed. FCBP must have a negative serum pregnancy test at screening.
* Able to adhere to the study visit schedule and other protocol requirements.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, uncontrolled intercurrent illness, or psychiatric illness/social condition that would prevent study participation.
* Concurrent use of any other anti-cancer agents or treatments or any other investigational agents.
* Treatment with strong CYP3A4/5 and/or CYP2D6 inhibitors
* Prior exposure to ibrutinib or ulocuplumab
* With the exception of low-dose aspirin, subjects enrolled in this study should not take concomitant medications that durably inhibit platelet function including marine oil tablets. For such medications a wash-out period of ≥ 7 days is required prior to starting treatment. Agents which inhibit platelet function transiently or inhibit coagulation by other mechanisms are restricted (e.g. use with caution). Medications that directly and durably inhibit platelet function include aspirin containing combinations, clopidogrel, dipyridamole, tirofiban, epoprostenol, eptifibatide, cilostazol, abciximab, ticlopidine, cilostazol.
* Participants should not take drugs that directly and durably inhibit coagulation with the exception of warfarin (coumadin) and heparin including low-molecular-weight heparin (LMWH), including enoxaparin, tinzaparin, etc.
* Any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Known CNS lymphoma.
* New York Heart Association classification III or IV heart failure.
* Known history of Human Immunodeficiency Virus (HIV), active infection with Hepatitis B Virus (HBV), and/or Hepatitis C Virus (HCV).
* Lactating or pregnant women.
* Grade > 2 toxicity (other than alopecia) continuing from prior anti-cancer therapy.
* Inability to swallow capsules
* History of non-compliance to medical regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P. Treon, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kipps TJ. Mining the Microenvironment for Therapeutic Targets in Chronic Lymphocytic Leukemia. Cancer J. 2021 Jul-Aug 01;27(4):306-313. doi: 10.1097/PPO.0000000000000536. PMID 34398557
- [Derived] Treon SP, Meid K, Hunter ZR, Flynn CA, Sarosiek SR, Leventoff CR, White TP, Cao Y, Roccaro AM, Sacco A, Demos MG, Guerrera ML, Kofides A, Liu X, Xu L, Patterson CJ, Munshi M, Tsakmaklis N, Yang G, Ghobrial IM, Branagan AR, Castillo JJ. Phase 1 study of ibrutinib and the CXCR4 antagonist ulocuplumab in CXCR4-mutated Waldenstrom macroglobulinemia. Blood. 2021 Oct 28;138(17):1535-1539. doi: 10.1182/blood.2021012953. PMID 34289017

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Level 1: Ibrutinib + Ulocuplumab 400mg Cycle 1 and 800mg Cycles 2-6: * Ibrutinib administered orally once daily for 48 cycles
  * Ulocuplumab administered intravenously at 400mg for Cycle 1 on Days 1, 8, 15, and 22. Ulocuplumab administered IV at 800mg for Cycles 2-6 on Days 1 and 15.
  Ulocuplumab: Ulocuplumab is a type of protein called an antibody that attacks CXCR4
  Ibrutinib: Ibrutinib small-molecule inhibitor of Bruton's tyrosine kinase (BTK) with potential antineoplastic activity
- Phase 1 Dose Level 2: Ibrutinib + Ulocuplumab 800 mg Cycle 1 and 1200mg Cycles 2-6: * Ibrutinib administered orally once daily for 48 cycles
  * Ulocuplumab administered intravenously at 800mg for Cycle 1 on Days 1, 8, 15, and 22. Ulocuplumab administered IV at 1200mg for Cycles 2-6 on Days 1 and 15.
  Ulocuplumab: Ulocuplumab is a type of protein called an antibody that attacks CXCR4
  Ibrutinib: Ibrutinib small-molecule inhibitor of Bruton's tyrosine kinase (BTK) with potential antineoplastic activity
- Phase 1 Dose Level 3: Ibrutinib + Ulocuplumab 800mg Cycle 1 and 1600mg Cycles 2-6: * Ibrutinib administered orally once daily for 48 cycles
  * Ulocuplumab administered intravenously at 800mg for Cycle 1 on Days 1, 8, 15, and 22. Ulocuplumab administered IV at 1600mg for Cycles 2-6 on Days 1 and 15.
  Ulocuplumab: Ulocuplumab is a type of protein called an antibody that attacks CXCR4
  Ibrutinib: Ibrutinib small-molecule inhibitor of Bruton's tyrosine kinase (BTK) with potential antineoplastic activity
Period: Overall Study
Arm/Group | Phase 1 Dose Level 1: Ibrutinib + Ulocuplumab 400mg Cycle 1 and 800mg Cycles 2-6 | Phase 1 Dose Level 2: Ibrutinib + Ulocuplumab 800 mg Cycle 1 and 1200mg Cycles 2-6 | Phase 1 Dose Level 3: Ibrutinib + Ulocuplumab 800mg Cycle 1 and 1600mg Cycles 2-6
Started | 7 | 3 | 3
Completed | 2 | 1 | 0
Not Completed | 5 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Study early termination by Sponsor | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 Dose Level 2: Ibrutinib + Ulocuplumab 800 mg Cycle 1 and 1200mg Cycles 2-6: * Ibrutinib administered orally once daily for 48 cycles
  * Ulocuplumab administered intravenously at 800mg for Cycle 1 on Days 1, 8, 15, and 22. Ulocuplumab administered IV at 1200mg for Cycles 2-6 on Days 1 and 15.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1: Ibrutinib + Ulocuplumab 400mg Cycle 1 and 800mg Cycles 2-6 | Phase 1 Dose Level 2: Ibrutinib + Ulocuplumab 800 mg Cycle 1 and 1200mg Cycles 2-6 | Phase 1 Dose Level 3: Ibrutinib + Ulocuplumab 800mg Cycle 1 and 1600mg Cycles 2-6 | Total
Number analyzed (Participants) | 7 | 3 | 3 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 3 | 11
  >=65 years | 1 | 1 | 0 | 2
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 70] | 63 [62 to 76] | 54 [53 to 64] | 61 [40 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 5 | 1 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 3 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 3 | 3 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 3 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Ulocuplumab
Description: MTD was determined by testing increasing doses up to 1600mg of ulocuplumab on dose escalation levels 1 to 3 with 3 to 7 participants each. MTD reflects the highest dose of ulocuplumab that did not cause a Dose-Limiting Toxicity (DLT) in >33% of participants. DLTs were defined as any Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE 4.0) grade 4 or 5 hematologic toxicities (anemia, neutropenia, or thrombocytopenia) and grade 3 or above non-hematologic toxicities. Exceptions were allowed for toxicities attributed to underlying disease, grade 3 infection, and easily reversible asymptomatic laboratory abnormalities, and nausea, vomiting, or diarrhea controlled by medications.
Time Frame: Up to 8 weeks for each dose level
Measure: Number; unit: milligram
Groups:
- All Participants: All participants who received at least 1 dose of Ulocuplumab, either at 400mg for cycle 1 and 800mg for cycle 2+, 800mg for cycle 1 and 1200mg for cycle 2+, or 800mg for cycle 1 and 1600mg for cycle 2+
Arm/Group | All Participants
Number analyzed (Participants) | 13
milligram | 1600

2. Secondary Outcome: Time to Minor Response
Description: Time in months to >25%-50% reduction in serum IgM from baseline
Time Frame: Response evaluated at each cycle day 1, starting at Cycle 2 Day 1 through Cycle 48
Population: All participants who received at least 1 dose of Ulocuplumab, either at 400mg for cycle 1 and 800mg for cycle 2+, 800mg for cycle 1 and 1200mg for cycle 2+, or 800mg for cycle 1 and 1600mg for cycle 2+
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1 Dose Level 1: Ibrutinib + Ulocuplumab 400mg Cycle 1 and 800mg Cycles 2-6 | Phase 1 Dose Level 2: Ibrutinib + Ulocuplumab 800 mg Cycle 1 and 1200mg Cycles 2-6 | Phase 1 Dose Level 3: Ibrutinib + Ulocuplumab 800mg Cycle 1 and 1600mg Cycles 2-6
Number analyzed (Participants) | 7 | 3 | 3
months | 1 [1 to 2] | 1 [1 to 1] | 1 [1 to 2]

3. Secondary Outcome: Time to Major Response
Description: Time in months to >50-90% reduction in serum IgM from baseline
Time Frame: Response evaluated at each cycle day 1, starting at Cycle 2 Day 1 through Cycle 48
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1 Dose Level 1: Ibrutinib + Ulocuplumab 400mg Cycle 1 and 800mg Cycles 2-6 | Phase 1 Dose Level 2: Ibrutinib + Ulocuplumab 800 mg Cycle 1 and 1200mg Cycles 2-6 | Phase 1 Dose Level 3: Ibrutinib + Ulocuplumab 800mg Cycle 1 and 1600mg Cycles 2-6
Number analyzed (Participants) | 7 | 3 | 3
months | 3 [1 to 4] | 1 [1 to 1] | 1 [1 to 3]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Time in months until >25% increase in serum IgM from nadir
Time Frame: Response and progression status evaluated at each cycle day 1, starting at Cycle 2 Day 1 through Cycle 48, and every 12 weeks during follow-up for up to 2 years after end of treatment
Population: Of the 13 participants enrolled, only 1 participant confirmed disease progression during the study period. Median PFS was not reached. The median follow-up time before participants follow-up was terminated for each participant is reported.
Measure: Median (Full Range); unit: months
Groups:
- Phase 1 Dose Level 2: Ibrutinib + Ulocuplumab 800 mg Cycle 1 and 1200mg Cycles 2-6: * Ibrutinib administered orally once daily for 48 cycles
  * Ulocuplumab administered intravenously at 400mg for Cycle 1 on Days 1, 8, 15, and 22. Ulocuplumab administered IV at 800mg for Cycles 2-6 on Days 1 and 15.
- Phase 1 Dose Level 3: Ibrutinib + Ulocuplumab 800mg Cycle 1 and 1600mg Cycles 2-6: * Ibrutinib administered orally once daily for 48 cycles
  * Ulocuplumab administered intravenously at 800mg for Cycle 1 on Days 1, 8, 15, and 22. Ulocuplumab administered IV at 1200mg for Cycles 2-6 on Days 1 and 15.
Arm/Group | Phase 1 Dose Level 1: Ibrutinib + Ulocuplumab 400mg Cycle 1 and 800mg Cycles 2-6 | Phase 1 Dose Level 2: Ibrutinib + Ulocuplumab 800 mg Cycle 1 and 1200mg Cycles 2-6 | Phase 1 Dose Level 3: Ibrutinib + Ulocuplumab 800mg Cycle 1 and 1600mg Cycles 2-6
Number analyzed (Participants) | 7 | 3 | 3
months | 20 [3 to 45] | 43 [35 to 44] | 37 [15 to 42]

ADVERSE EVENTS:
Time Frame: Adverse events were captured after treatment initiation and through 30 days of the last dose, up to 4 years.
Arm/Group | Phase 1 Dose Level 1: Ibrutinib + Ulocuplumab 400mg Cycle 1 and 800mg Cycles 2-6 | Phase 1 Dose Level 2: Ibrutinib + Ulocuplumab 800 mg Cycle 1 and 1200mg Cycles 2-6 | Phase 1 Dose Level 3: Ibrutinib + Ulocuplumab 800mg Cycle 1 and 1600mg Cycles 2-6
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/7 | 1/3 | 1/3
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1: Ibrutinib + Ulocuplumab 400mg Cycle 1 and 800mg Cycles 2-6 (N=7) | Phase 1 Dose Level 2: Ibrutinib + Ulocuplumab 800 mg Cycle 1 and 1200mg Cycles 2-6 (N=3) | Phase 1 Dose Level 3: Ibrutinib + Ulocuplumab 800mg Cycle 1 and 1600mg Cycles 2-6 (N=3)
Brain injury from motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1: Ibrutinib + Ulocuplumab 400mg Cycle 1 and 800mg Cycles 2-6 (N=7) | Phase 1 Dose Level 2: Ibrutinib + Ulocuplumab 800 mg Cycle 1 and 1200mg Cycles 2-6 (N=3) | Phase 1 Dose Level 3: Ibrutinib + Ulocuplumab 800mg Cycle 1 and 1600mg Cycles 2-6 (N=3)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 0 (0)
Bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Heart racing (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear bleeding (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear granuloma (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Corneal ulcer (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chelitiis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Blood blisters (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (2) | 1 (1)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0)
Hair growing faster (General disorders) | 0 (0) | 0 (0) | 1 (1)
Heavy legs (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Sciatica (General disorders) | 1 (1) | 0 (0) | 0 (0)
Temperature sensitivity (General disorders) | 0 (0) | 0 (0) | 1 (1)
Tympanic membrane perforation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 4 (4) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tick bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 6 (6) | 3 (3) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2)
Headache (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Jittery (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth numbness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Irregular Menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Blood blisters (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Boil (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Irregular mole (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Onychoschizia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash NOS (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Stye (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT03225716/Prot_SAP_000.pdf